CLINICAL TRIAL: NCT04017858
Title: PARQVE Prior to Total Knee Replacement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Marcia Uchoa Rezende, Full Professor in Orthopedics and Traumatology, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04019418.7.0000.0068
Record Dates: First submitted 2019-06-26; First posted 2019-07-12 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Knee Osteoarthritis
Keywords: Total knee arthroplasty; Exercise; Preoperative; Complications
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Multiprofessional and educational Program prior to Total knee replacement TKA. (PARQVE TKA).
  Interventions: Behavioral: Multiprofessional and educational Program prior to Total knee replacement TKA. (PARQVE TKA).
- Control (Active Comparator): Patients will be submitted to total knee replacement.
  Interventions: Behavioral: Patients will be submitted to total knee replacement.

INTERVENTIONS:
Behavioral: Multiprofessional and educational Program prior to Total knee replacement TKA. (PARQVE TKA). — Patients will participate in two days of about knee OA lectures two months apart, will also come to the hospital at months 1, 3 and 5 after the first class to consult about nutritional habits; at months 4 and 6 to participate in a group therapy session with the psychologists, 7 sessions with the physical therapy followed by 7 sessions with the physical educators team. Following this program, patients will be operated (total knee arthroplasty).
  Answer Womac, VAS, Lequesne, BMI and body fat percentage - at inclusion, one week prior to surgery, 1 and 6 months postoperatively.
  Days of hospital stay will be measured by the number of nights the patients stay in the hospital postoperatively and also days in semi-intensive.
  Minutes and type of physical activity - Answer at inclusion and six months postoperatively.
  Perform STS30 and TUG at inclusion, one week prior to surgery, 1 and 6 months postoperatively Costs will be evaluated for cost-effectiveness and cost-utility analysis
  Arms: Experimental
Behavioral: Patients will be submitted to total knee replacement. — Patients will be submitted to total knee replacement, without Multiprofessional and educational Program Answer Womac, VAS, Lequesne, BMI and body fat percentage - at inclusion, one week prior to surgery, 1 and 6 months postoperatively.
  Days of hospital stay will be measured by the number of nights the patients stay in the hospital postoperatively and also days in semi-intensive.
  Minutes and type of physical activity - Answer at inclusion and six months postoperatively.
  Perform the STS30 and TUG at inclusion, one week prior to surgery, 1 and 6 months postoperatively
  Arms: Control

SUMMARY:
Introduction: Elderly patients, the majority of the population submitted to total knee arthroplasty (TKA), have a lower capacity for adaptation to hospitalization and surgical stress. Exercise before cardiac and abdominal elective surgery was shown to reduce the number of complications. Studies have shown that preoperative exercise improves functional performance, strength and may decrease hospital stay after an ATJ. Objective: To evaluate if the program exercises before TKA improves quality of life, function, pain and body composition, time of hospitalization and number of complications of patients submitted to TKA. Methods: 44 patients awaiting TKA in IOT-HC-FMUSP will be divided into two groups. Half of the patients will undergo a multiprofessional and physical activity educational program for 20 weeks while the other half will wait for the TCA in the outpatient clinic. Patients will be evaluated through functional tests (sit-up and 30-second tests and time up and go), standardized questionnaires (WOMAC and Lequesne), quality of life scales (Euroqol-EQ-5D-5L), pain (through VAS), body composition and bone density (through densitometry), time of hospitalization and complications resulting from TKA. All of the above parameters will be assessed at baseline and 1 and 6 months after TKA. All project costs will be reported and a cost-effectiveness and cost-utility analysis will be performed.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is generally advocated as an effective operation to alleviate symptoms in people suffering from knee osteoarthritis (OAJ). Such statements are often made from a medical and biomechanical perspective (in terms of low complication rates and prosthesis failure) instead of the patient's perspective (pain and functional outcome). Hawker et al. Demonstrated that almost half of the patients submitted to TKA had poor results regarding pain and function; these were mainly elderly patients with additional comorbidities.

Elderly patients, a majority of the population submitted to TKA, have a lower capacity for adaptation to hospitalization and surgical stress. Exercise before cardiac and abdominal elective surgery was shown to reduce the number of complications.

Pre- and postoperative physical therapy may increase the functional recovery of patients undergoing TKA. To date, a number of reviews have been available that demonstrate that preoperative exercise in subjects awaiting TKA has little value in postoperative outcomes. However, most of the included studies investigated the efficacy of preoperative exercise in generally healthy adults, while, in essence, eligible individuals with comorbidities and / or elderly were excluded. Therefore, to understand and appreciate the true potential of preoperative therapeutic exercise, the investigators needs to evaluate studies that included individuals at highest risk for disappointing outcomes after surgery. Two studies are available that investigated the merits of preoperative exercise in patients with increased risk of late functional recovery or increased length of hospital stay. Topp et al. investigated the efficacy of the therapeutic exercise in patients with low preoperative functional level pending TKA. This study demonstrated that, after 3 months, the functional performance level and strength of the preoperative exercise group was greater than the control group. Hansen et al. have demonstrated that, in the context of FAST TRACK, the preoperative therapeutic exercise in individuals with a higher risk of delayed recovery may further decrease hospital stay (one additional day) after TKA.

Even excluding patients with comorbidities Villadsen et al. demonstrated that patients undergoing an exercise program before TKA recovered faster after surgery.

In previous work performed by the authors, patients submitted to an education and physical activity program showed improvement in WOMAC, which can be reproduced in any basic health care unit.

Thus the investigators believe that the sum of an education program associated with preoperative exercises needs to be considered as a tool to help recovery after TKA, as it is an inexpensive, well tolerated and easily implemented intervention in UBS.

ELIGIBILITY:
Inclusion Criteria:

* Men and women diagnosed with OAK with comorbidities (metabolic syndrome, i.e. OAK + at least two overweight / central obesity, diabetes, dyslipidemia, hypertension)
* Age between 60 and 75 years who are waiting Total knee arthroplasty
* Patients not submitted to previous arthroplasty in the lower limbs.
* Patients not submitted to infiltration in the knees up to 6 months before the study.
* Patients with no personal history of cognitive, psychiatric and / or neurological disorders, whose symptoms presented at the time of evaluation are related or significantly interfere with the functions of attention, memory, logical reasoning, comprehension, in order to impair the assimilation of the given guidelines.
* Patients with no personal history of inflammatory arthritis (rheumatoid arthritis, for example)
* Patients able to read, understand and respond to questionnaires and perform functional tests.

Exclusion Criteria:

* Missing in interventions and do not perform the tasks determined by the professionals.
* Patients submitted to infiltration in the knees during the study.
* Patients diagnosed with chronic inflammatory arthritis (rheumatoid arthritis, for example) during the study.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2019-10-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Change the functional results of patients in the sit to stand 30 seconds | 6 months
  To evaluate whether the multiprofessional treatment program and exercises improves the functional results of patients in the sit to stand 30 seconds (STS30) in the 6th. month of the study (Project PARQVE prior to TKA).

SECONDARY OUTCOMES:
Improves results of Sit to Stand 30 Seconds Test | 1 month
  Perform Sit to Stand 30 Seconds Test - Involves recording the number of stands a person can complete in 30 seconds, more fast better.
Improves results of Time Up and Go Test | 1 month and 6 months
  Perform Time Up and Go Test - The time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down, faster perform better.
Improves results of Womac Questionnaire | 1 month and 6 months
  Answer Womac Questionnaire - Ranges: minimum 0 (Better, no pain and limitation) / maximum 96 (Worst pain and limitation)
Improves results of Lequesne Questionnaire | 1 month and 6 months
  Answer Lequesne Questionnaire - Ranges: minimum 0 (Better, no limitation) / maximum 24 (Worst limitation)
Improves results of Visual Analogue Scale | 1 month and 6 months
  Answer Visual Analogue Scale - Ranges: minimum 0 (Better, no pain) / maximum 100 (Worst pain)
Improves results of EuroQol Scale | 1 month and 6 months
  Answer EuroQol Scale - Ranges: minimum 0 (Better) / maximum 2 (Worst)
Increases lean mass percentage | 1 month and 6 months
  Calculate lean mass
Decreases fat percentage | 1 month and 6 months
  Calculate fat percentage
Increases minutes per week of physical activity | 6 months
  Answer questionnaire

OTHER OUTCOMES:
Decreases length of hospital stay | 6 months
  Make an economic evaluation of the program regarding cost-effectiveness and cost-utility.

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme P Ocampos, MD, Principal Investigator — University of São Paulo General Hospital
Locations (1):
- Instituto de Ortopedia e Traumatologia do Hospital das Clinicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hawker GA, Badley EM, Borkhoff CM, Croxford R, Davis AM, Dunn S, Gignac MA, Jaglal SB, Kreder HJ, Sale JE. Which patients are most likely to benefit from total joint arthroplasty? Arthritis Rheum. 2013 May;65(5):1243-52. doi: 10.1002/art.37901. PMID 23459843
- [Background] Hoogeboom TJ, Dronkers JJ, Hulzebos EH, van Meeteren NL. Merits of exercise therapy before and after major surgery. Curr Opin Anaesthesiol. 2014 Apr;27(2):161-6. doi: 10.1097/ACO.0000000000000062. PMID 24500337
- [Background] Mak JC, Fransen M, Jennings M, March L, Mittal R, Harris IA; National Health and Medical Research Council (NHMRC) of Australia. Evidence-based review for patients undergoing elective hip and knee replacement. ANZ J Surg. 2014 Jan-Feb;84(1-2):17-24. doi: 10.1111/ans.12109. Epub 2013 Mar 15. PMID 23496209
- [Background] Hoogeboom TJ, Oosting E, Vriezekolk JE, Veenhof C, Siemonsma PC, de Bie RA, van den Ende CH, van Meeteren NL. Therapeutic validity and effectiveness of preoperative exercise on functional recovery after joint replacement: a systematic review and meta-analysis. PLoS One. 2012;7(5):e38031. doi: 10.1371/journal.pone.0038031. Epub 2012 May 31. PMID 22675429
- [Background] Topp R, Swank AM, Quesada PM, Nyland J, Malkani A. The effect of prehabilitation exercise on strength and functioning after total knee arthroplasty. PM R. 2009 Aug;1(8):729-35. doi: 10.1016/j.pmrj.2009.06.003. PMID 19695525
- [Background] Hansen TB, Bredtoft HK, Larsen K. Preoperative physical optimization in fast-track hip and knee arthroplasty. Dan Med J. 2012 Feb;59(2):A4381. PMID 22293051
- [Background] Villadsen A, Overgaard S, Holsgaard-Larsen A, Christensen R, Roos EM. Postoperative effects of neuromuscular exercise prior to hip or knee arthroplasty: a randomised controlled trial. Ann Rheum Dis. 2014 Jun;73(6):1130-7. doi: 10.1136/annrheumdis-2012-203135. Epub 2013 May 9. PMID 23661494
- [Background] Wright AA, Cook CE, Baxter GD, Dockerty JD, Abbott JH. A comparison of 3 methodological approaches to defining major clinically important improvement of 4 performance measures in patients with hip osteoarthritis. J Orthop Sports Phys Ther. 2011 May;41(5):319-27. doi: 10.2519/jospt.2011.3515. Epub 2011 Feb 18. PMID 21335930